CLINICAL TRIAL: NCT04217707
Title: Mental and Physical Health Benefits of Pre- and Post-Surgical Transgender Therapeutic Support Groups
Brief Title: Transgender Therapeutic Support Groups
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study unable to be conducted due to COVID.
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Rachel Narr, Postdoctoral Fellow, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0001
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Gender Dysphoria in Adolescents and Adults
MeSH Terms: interventions — Lead

STUDY DESIGN:
Intervention Model Description: Participants will be patients drawn from already-existing therapeutic support groups for transgender patients who are hoping to undergo or have undergone gender-affirming surgeries. Research participants will participate in the groups as usual, and after each of their first eight attended sessions, will be asked to fill out outcomes of interest again. Due to the possibility that participants may not attend eight group sessions, length of time for them to attend eight sessions will be capped at 6 months, and participants will be asked to fill out measures again at six months following their enrollment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre- and Post-Surgical Transgender Therapeutic Support Groups (Other)
  Interventions: Behavioral: Pre- and Post-Surgical Transgender Therapeutic Support Group

INTERVENTIONS:
Behavioral: Pre- and Post-Surgical Transgender Therapeutic Support Group — Participants will be patients drawn from already-existing therapeutic support groups for transgender patients who are hoping to undergo or have undergone gender-affirming surgeries. Participants will be assured that there will be no changes to their care or decisions about their surgeries if they elect not to participate in the research portion of the groups, but would still like to attend groups as a non-research participant. Prior to their first group session, participants will be arrive early to go over consent again and allow participants to sign the consent form and fill out baseline measures of the outcomes of interest. Following this, research participants will participate in the groups as usual, and after each of their first 8 attended sessions, will be asked to fill out outcomes of interest again. Length of time for them to attend 8 sessions will be capped at 6 months, and participants will be asked to fill out measures again at six months following their enrollment.

SUMMARY:
This study seeks to explore the effects for transgender people undergoing surgical interventions of participating in pre/post-surgical therapeutic support groups in order to assess the value of adding these programs to hospital systems that are offering gender-affirming surgeries. Participation in either therapeutic support group is expected to increase subjective well-being, increase perceived social support, and decrease clinically significant mental health symptoms compared to participants' baseline scores. It is expected that perceived social support will mediate the relation between group participation and improved subject well-being and mental health scores. In addition, participation in the post-surgical therapeutic support group is expected to reduce the average number of emergency department visits for participants in the group compared with transgender patients, post-gender-affirming surgery, in the hospital as a whole.

DETAILED DESCRIPTION:
At present, in the scientific literature, there are no known studies of the effectiveness of therapeutic support groups for supporting mental and physical health in transgender or gender nonconforming (TGNC)-identified individuals who are undergoing gender-affirming surgical interventions. Gender affirmation surgeries have been shown to decrease anxiety and depression, and increase well-being for TGNC individuals compared to the well-being of TGNC individuals who do not access surgery. In spite of this, surgery is inherently stressful for people undergoing it, and there are a plethora of medical and psychological complications that may be faced by people undergoing these surgeries.

Denver Health has greatly expanded gender-affirming interventions in the past three years due to the creation of the Center of Excellence; however, mental health services are still catching up. While support from other TGNC individuals has proven to be effective in general for reducing anxiety and depression, and community support groups have begun to be offered more regularly to support TGNC individuals, surgical support groups appear to largely not be offered. However, a high proportion of TGNC individuals express a desire for post-surgical support around surgery results (84.6% in a sample of 415 people), and over 90% of people are in favor of peer support around medical interventions more broadly. In other areas, specifically bariatric surgery, peer therapeutic support groups have been found to help with continued post-operative weight loss and mental health, likely due to the additional opportunities for support and connection with others undergoing similar things, group provision of ideas, and additional therapeutic support. While individual therapy is, and should continue to be, offered for this population, the addition of a group attended by individuals going through similar situations is likely to be helpful above and beyond individual therapy due to the provision of peer support, as well as the opportunity for participants to offer support to their peers. Seeing oneself as a help provider, rather than simply a help recipient (helper-therapy principle) has been demonstrated to have a powerful impact on the helper's own well-being across a host of medical and psychological situations.

Currently, therapeutic support groups are being developed to be offered to TGNC patients at Denver Health who are undergoing gender-affirming surgeries. Investigators will systematically collect data on well-being and mental health, as well as the mediating effect of feelings of cohesion on well-being, as well as the number of emergency department visits for participants in the groups as compared to the average number of emergency department visits across all TGNC patients in the Denver Health system for patients involved in these groups. Given the deficit of groups of this nature, as well as information on the helpfulness of therapeutic support groups for people undergoing gender-affirming surgeries, the investigators expect that this may be the first study on this topic. The study hypothesis is that participants in pre- and post-surgical support groups will experience increased well-being and mental health over a six month period, and that these increases will be mediated by group cohesion. Investigators also expect that attendance at these groups will lead to lower utilization of emergency services due to decreased anxiety and distress.

ELIGIBILITY:
Inclusion Criteria:

* Transgender and gender non-conforming adults who take part in therapeutic support groups aimed at patients prior to and after gender-affirming surgical interventions.

Exclusion Criteria:

* Age < 18
* Substance abuse as primary presenting problem and unable to maintain sobriety for group
* Severe mental illness with acute psychosis or paranoia
* Patients with a very high need for crisis management
* Patients with diagnosis of Antisocial Personality Disorder
* Patients with severe cognitive impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender-identified individuals
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Well-Being | Up to 6 months
  Subjective well-being will be assessed with the Short Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS). This is a 7-item scale assessing different aspects of mental well-being over the previous two weeks. It is scored on a 5-point Likert scale ranging from "None of the time" to "All of the time." The SWEMWBS has excellent internal consistency (Cronbach's α = .90), has shown both strong convergent and divergent validity, and has been validated in multiple populations and languages. In addition, this scale has been demonstrated to be sensitive to change over time in clinical populations receiving therapeutic intervention.
Broad mental health symptoms | Up to 6 months
  Broad mental health symptoms will be measured with the Mental Health Inventory - 5, which is a 5-item measure of general mental health symptoms over the past month. Symptoms assessed include symptoms characteristic of depression and anxiety in particular. Cronbach's α for this scale = .84, and it demonstrates good construct and convergent validity. In addition, this measure has been demonstrated to be sensitive to levels of social support.
Perceived social support | Up to 6 months
  Perceived social support will be evaluated using the 8-item Perceived Support subscale from the Berlin Social Support Scales. This subscale covers both emotional and instrumental support, focusing on how much support the respondents perceive themselves to be likely to receive, which has been shown to more strongly correlate with mood, adjustment, and wellness than objectively-measured received support. Each individual scale has been assessed in addition to the full measure, and the Perceived Support subscale has been found to have good internal consistency (Cronbach's α = .83. In addition, this measure has been shown to be sensitive to change in clinical populations.

SECONDARY OUTCOMES:
Emergency department visits | 6 months
  Emergency department visits following surgery over a six-month period will be assessed using patient medical charts. Average number of visits by study participants will be compared to average number of visits by all transgender patients in our hospital system undergoing gender-affirming surgeries. Comparison emergency department visits will not be linked with and individuals or protected health information (PHI), and will be an average across all patients in this demographic group.

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branstrom R, Pachankis JE. Reduction in Mental Health Treatment Utilization Among Transgender Individuals After Gender-Affirming Surgeries: A Total Population Study. Am J Psychiatry. 2020 Aug 1;177(8):727-734. doi: 10.1176/appi.ajp.2019.19010080. Epub 2019 Oct 4. PMID 31581798
- [Background] Pflum, S.R., Testa, R.J., Balsam, K.F., Goldblum, P.B., & Bongar, B. (2015). Social support, trans community connectedness, and mental health symptoms among transgender and gender nonconforming adults. Psychology of Sexual Orientation and Gender Identity, 2(3), 281-286.
- [Background] Eyssel J, Koehler A, Dekker A, Sehner S, Nieder TO. Needs and concerns of transgender individuals regarding interdisciplinary transgender healthcare: A non-clinical online survey. PLoS One. 2017 Aug 28;12(8):e0183014. doi: 10.1371/journal.pone.0183014. eCollection 2017. PMID 28846715
- [Background] Huberman, W.L. (2008). One psychologist's 7-year experience in working with surgical weight loss: The role of the mental health professional. Primary Psychiatry, 15(8), 42-47.
- [Background] Livhits M, Mercado C, Yermilov I, Parikh JA, Dutson E, Mehran A, Ko CY, Shekelle PG, Gibbons MM. Is social support associated with greater weight loss after bariatric surgery?: a systematic review. Obes Rev. 2011 Feb;12(2):142-8. doi: 10.1111/j.1467-789X.2010.00720.x. PMID 20158617
- [Background] Riessman, F. (1965). The "helper" therapy principle. Social Work, 10(2), 27-32.
- [Background] Weinstein N, Ryan RM. When helping helps: autonomous motivation for prosocial behavior and its influence on well-being for the helper and recipient. J Pers Soc Psychol. 2010 Feb;98(2):222-44. doi: 10.1037/a0016984. PMID 20085397
- [Background] Hutchinson DS, Anthony WA, Ashcraft L, Johnson E, Dunn EC, Lyass A, Rogers ES. The personal and vocational impact of training and employing people with psychiatric disabilities as providers. Psychiatr Rehabil J. 2006 Winter;29(3):205-13. doi: 10.2975/29.2006.205.213. PMID 16450932
- [Background] Pagano ME, Post SG, Johnson SM. Alcoholics Anonymous-Related Helping and the Helper Therapy Principle. Alcohol Treat Q. 2010 Jan 1;29(1):23-34. doi: 10.1080/07347324.2011.538320. Epub 2011 Jan 19. PMID 23525280
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Ng Fat L, Scholes S, Boniface S, Mindell J, Stewart-Brown S. Evaluating and establishing national norms for mental wellbeing using the short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS): findings from the Health Survey for England. Qual Life Res. 2017 May;26(5):1129-1144. doi: 10.1007/s11136-016-1454-8. Epub 2016 Nov 16. PMID 27853963
- [Background] Shah N, Cader M, Andrews WP, Wijesekera D, Stewart-Brown SL. Responsiveness of the Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS): evaluation a clinical sample. Health Qual Life Outcomes. 2018 Dec 22;16(1):239. doi: 10.1186/s12955-018-1060-2. PMID 30577856
- [Background] Vaingankar JA, Abdin E, Chong SA, Sambasivam R, Seow E, Jeyagurunathan A, Picco L, Stewart-Brown S, Subramaniam M. Psychometric properties of the short Warwick Edinburgh mental well-being scale (SWEMWBS) in service users with schizophrenia, depression and anxiety spectrum disorders. Health Qual Life Outcomes. 2017 Aug 1;15(1):153. doi: 10.1186/s12955-017-0728-3. PMID 28764770
- [Background] Schwarzer, R. & Schulz, U. (2013). Berlin Social Support Scales (BSSS). Measurement Instrument Database for the Social Science. Retrieved from www.midss.ie
- [Background] Norris FH, Kaniasty K. Received and perceived social support in times of stress: a test of the social support deterioration deterrence model. J Pers Soc Psychol. 1996 Sep;71(3):498-511. doi: 10.1037//0022-3514.71.3.498. PMID 8831159
- [Background] Wethington E, Kessler RC. Perceived support, received support, and adjustment to stressful life events. J Health Soc Behav. 1986 Mar;27(1):78-89. No abstract available. PMID 3711634
- [Background] McCabe CJ, Thomas KJ, Brazier JE, Coleman P. Measuring the mental health status of a population: a comparison of the GHQ-12 and the SF-36 (MHI-5). Br J Psychiatry. 1996 Oct;169(4):516-21. doi: 10.1192/bjp.169.4.516. PMID 8894205
- [Background] Ware, J., Kosinki, M., & Gandek, B. (2000). SF-36 health survey: Manual & Interpretation Guide. Lincoln: Quality Metric Incorporated.